CLINICAL TRIAL: NCT02363400
Title: Phase III Randomized Trial of Immediate Adjuvant Chemotherapy or Delayed Salvage Chemotherapy in Nasopharyngeal Carcinoma Patients With Post-radiation Detectable Plasma EBV DNA
Brief Title: A Phase III Trial in NPC With Post-radiation Detectable Plasma EBV DNA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting progress behind expectation
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Mackay Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Taichung Veterans General Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1313
Record Dates: First submitted 2014-12-04; First posted 2015-02-16 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2016-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma (NPC); Epstein-Barr virus (EBV); radiotherapy (RT); Plasma EBV DNA(pEBV DNA); Adjuvant Chemotherapy; PET-CT scan at Pre-Tx restaging
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Epirubicin; Cisplatin; Tegafur; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Chemotherapy (Experimental): MEP followed by oral Tegafur-uracil
  Interventions: Drug: MEP
- control arm (No Intervention): closely followed with frequency similar to the experiemental arm

INTERVENTIONS:
Drug: MEP — Adjuvant Chemotherapy
  Other Names: epirubicin; cisplatin; oral Tegafur-uracil; mitomycin-C
  Arms: Adjuvant Chemotherapy

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a geographically endemic, Epstein-Barr virus (EBV)-associated carcinoma of epidermoid origin. It occurs most commonly in Southern China and Southeast Asia. The NPC cells are poorly differentiated or undifferentiated with a high incidence of lymphatic and hematological dissemination. Because of the inherent anatomic constraints and a high degree of radiosensitivity, radiotherapy (RT) has been the primary treatment for NPC patients.

NPC is also a chemosensitive tumor. Various modes of combined chemoradiotherapy have been used to treat NPC patients with advanced-stage diseases during recent 20 years. However, treatment outcome for locoregionally advanced NPC is still unsatisfactory.

DETAILED DESCRIPTION:
The current NCCN guidelines recommend that CCRT + adjuvant chemotherapy for advanced (stage III-IV) NPC, originated from the results of the Intergroup study [69]. However, all meta-analysis reported no any benefit in using adjuvant chemotherapy for NPC patients [82-85]. These contradictions puzzle most oncologists for decades. In our opinion, routine delivery of post-radiation adjuvant chemotherapy after RT±induction/concurrent chemotherapy for "all" advanced-stage NPC patients should be re-considered. The major goal of adjuvant chemotherapy in NPC is to reduce the occurrences of distant failure. But, not all advanced NPC patients need adjuvant chemotherapy. In our previous phase III study, only 19.1% (27/141) NPC patients with 1988 AJCC stage III-IV disease developed distant failure after CCRT . In another study of 210 NPC patients with 1997 AJCC stage IIB-IVB treated by induction chemotherapy + RT, 55 patients (26.2%) suffered from subsequent distant metastasis [67]. We should remember that unnecessary adjuvant therapy is frequently used. For example, if the target patients have as high as 50% subsequent distant failure rate, and the adjuvant therapy protocol has a 50% control rate for the subclinical disease. When we treat all target patients, only 25% patients benefit from the adjuvant therapy because of unnecessary treatment in 50% and ineffective treatment in another 25% patients. Thus, adjuvant therapy should be designed for "selected" patients. For NPC patients, pEBV DNA-guided adjuvant therapy trial is very reasonable. We plan to prove that adjuvant chemotherapy is beneficial for post-radiation detectable pEBV DNA patients in this prospective multi-center trial. We will conduct another trial to investigate (compare) which adjuvant chemotherapy regimen is the best one in the future.

ELIGIBILITY:
Inclusion Criteria:

1.Histological proven NPC.

2.2010 AJCC stage II-IVB.

3.Age ≧ 20 years old.

4.Performance status of ECOG ≦ 2.

5.Finished RT ≧ 66 Gy (± induction and/or concurrent chemotherapy).

6.pEBV DNA > 0 copy/ml at 1±1 week post-RT.

7.Re-staging work-ups at 10±2 weeks post-RT showing no active lesions.

8.Adequate liver, renal, and bone marrow function 4 weeks before randomization.

9.Signed informed consent.

Exclusion Criteria:

1. Pathologically-proven the presence of locoregional disease and/or distant metastasis.
2. Unequivocally-shown active NPC (locoregional/distant) by imaging studies.
3. Inadequate RT.
4. Received any post-RT adjuvant chemotherapy.
5. pEBV DNA = 0 copy/ml at 1±1 week post-RT.
6. Previous delivery of cisplatin dose > 600 mg/m2.
7. Previous delivery of epirubicin > 360 mg/m2.
8. History of a malignancy except those treated with curative intent for skin cancer (other than melanoma), in situ cervical cancer, ductal carcinoma in situ (DCIS) of breast.
9. Severe cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the last 12 months; chronic obstructive pulmonary disease exacerbation other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders.
10. Female patients who are pregnant or lactating.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time to progression | 5 years

SECONDARY OUTCOMES:
Progression-free survival and relapse rate | 5 years
Overall survival | 5 years
Toxicity profile and tolerance, according to CTCAE 4.1 | 5 years
Predicting value of plasma EBV DNA | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ching Lin, MD, PHD, Study Chair — Taichung Veterans General Hospital; Tsang-Wu Liu, MD, Study Director — National Health Research Institutes, Taiwan; Jin-Ching Lin, MD, PhD, Principal Investigator — Taichung Veterans General Hospital; Yi-Fang Chang, MD, PhD, Principal Investigator — Mackay Memorial Hospital; Ching-Yun Hsieh, MD, Principal Investigator — China Medical University Hospital; Chia-Jui Yen Yen, MD. PhD, Principal Investigator — National Cheng-Kung University Hospital; Yaoh-Shiang Lin, MD, Principal Investigator — Kaohsiung Veterans General Hospital.; Stella Yu-Chen Tsai, MD, Principal Investigator — Sun Yat-sen University; Hsiao-Hui Tsou, PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (6):
- Taiwan (6):
  - Kaohsiung Veterans General Hospital., Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - Sun Yat-sen University, Taipei

IPD SHARING:
Plan to Share IPD: No